CLINICAL TRIAL: NCT00580008
Title: Evaluation Using CTA to Investigate and Detect Atherosclerotic Graft Disease (ELUCIDATE)
Brief Title: Evaluation Using Computed Tomography Angiography (CTA) to Investigate and Detect Atherosclerotic Graft Disease (ELUCIDATE)
Acronym: ELUCIDATE)
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Kavitha Chinnaiyan, Director, Cardiovascular Imaging Education, Corewell Health East
Other Study IDs: 2007-144
Record Dates: First submitted 2007-12-17; First posted 2007-12-24 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Arteriosclerosis of Coronary Artery Bypass Graft; Coronary Artery Disease
Keywords: tomography; coronary artery disease; coronary artery bypass grafting; vein graft
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum banking
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of clinical research is to look at the nature of disease and try to develop improved methods to diagnose and treat disease.The goal of this study is to evaluate the use of computed tomography (CT) scan of the heart in the diagnosis of disease in vein grafts after bypass surgery.

DETAILED DESCRIPTION:
Patients who have bypass surgery with using vein grafts from their legs (saphenous veins) have a very high risk of developing blockages in the grafts. It has been shown in previous studies that the progression of disease in vein grafts is very quick and can result in chest pain, heart attacks or death. In the past, evaluation of the grafts was possible with heart catheterization only. The technique of CT scan is currently considered an effective way to look at vein grafts as well as the arteries around the heart to identify blockages.

Certain blood proteins have been associated with rapid progression of vein graft blockages. Our purpose is to not only to identify blockages at different stages after bypass surgery, but to investigate the causes of the rapid progression of the disease, including clinical history, risk factors and the blood proteins.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent.
2. Age equal to or greater than 18 years.
3. One(-/+60days), 3 (-/+60days), 5 (-/+60days), or 7 (-/+60days) years after coronary artery bypass graft surgery.

Exclusion Criteria:

1. Renal (kidney) insufficiency (creatinine greater than or equal to 1.6) or renal (kidney) failure requiring dialysis.
2. Atrial fibrillation (type of heart rhythm) or other markedly irregular rhythm.
3. Inability or refusal to provide informed consent.
4. Pregnancy or unknown pregnancy status.
5. Age less than 18 years.
6. Clinical instability as deemed by the attending physician, including cardiogenic shock, hypotension (low blood pressure-systolic blood pressure less than 90 mmHg), refractory hypertension (high blood pressure) (systolic blood pressure greater than 180 mmHg), sustained ventricular or atrial arrhythmia (types of heart rhythm) requiring intravenous medications.
7. Inability to tolerate beta-blockers, including those with chronic obstructive pulmonary disease (temporary narrowing of the tubes in the lungs) (or asthma requiring maintenance inhaled bronchodilators or steroids, complete heart block (chambers in the heart not beating in sync), second-degree atrioventricular block (chambers in the heart not beating in sync).
8. Known contrast dye allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Referrals from physicians' office Patients' self-referral Age greater than 18 years old Both genders
Sampling Method: Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2007-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Morphological characteristics of vein grafts | two years
  To identify the presence of and morphological characteristics of vein graft disease in patients at 1 and 2 years post bypass surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Safian, MD, Principal Investigator — Corewell Health East; Kavitha Chinnaiyan, MD, Principal Investigator — Corewell Health East; Gil Raff, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States